Document: TDOC-0057261 Version: 2.0; Most-Recent; Effective; CURRENT

Status: Effective

#### **Short Title:**

## Statistical Analysis Plan CLY935-C008 / NCT04403542

#### **Full Title:**

## Statistical Analysis Plan CLY935-C008

Protocol Title: Pilot Clinical Performance of a Silicone Hydrogel Lens for Up to Six Nights of Extended Wear

Protocol TDOC Number: TDOC-0056933

Author:

**Approvals:** See last page for electronic approvals

Job Notes:

This is the first revision (Version 2.0) of the Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 2.0 of the study protocol.

Alcon - Business Use Only Statistical Analysis Plan

Version: 2.0; Most-Recent; Effective; CURRENT

Status: Effective

Executive Summary:

Key Objective:

The primary objective is to assess initial safety and performance of the soft contact lens when worn in an extended wear modality (ie, up to 6 nights/7 days of continuous wear) as compared to the BIOFINITY® soft contact lens (Biofinity).

Alcon - Business Use Only Statistical Analysis Plan

Effective Date: 21-Jul-2020 Version: 2.0; Most-Recent; Effective; CURRENT Document: TDOC-0057261

Status: Effective

#### **Table of Contents**

| Statistic | ıl Analysis Plan CLY935-C008 | ] |
|-----------|-----------------------------------------------------|-----|
| Table of | Contents | 2 |
| List of T | ables | |
| 1 | Study Objectives and Design | |
| 1.1 | Study Objectives | |
| 1.2 | Study Description | |
| 1.3 | Randomization. | |
| 1.4 | Masking | |
| 2 | Analysis Sets | 6 |
| 2.1 | Safety Analysis Set | 6 |
| 3 | Subject Characteristics and Study Conduct Summaries | |
| 4 | Effectiveness Analysis Strategy | |
| 4.3.1 | Primary Effectiveness Analyses | 8 |
| 5 | Safety Analysis Strategy | 1( |
| 5.1 | Safety Endpoints | 1( |
| 5.2 | Safety Hypotheses | 1( |
| 5.3 | Statistical Methods for Safety Analyses | 11 |
| 5.3.1 | Adverse Events | 11 |
| 5.3.2 | Biomicroscopy Findings | |
| 5.3.3 | Device Deficiencies | 12 |
| 7 | Sample Size and Dayyor Calculations | 1 4 |
| 7 | Sample Size and Power Calculations | 14 |

| | isiness Use Only Statistical Analysis Plan | |
|---|---|---|
| Document: T<br>Status: Effe | CDOC-0057261 Version: 2.0; Most-Recent; Effective | e; CURRENT |
| 8 | References | 12 |
| 9 | Revision History | 12 |
| 10 | Appendix | 14 |
| | List of Tables | |
| Table 1–1 | Study Description Summary | 5 |
| Table 10–1 | Overview of Study Plan | 14 |

Document: TDOC-0057261 Version: 2.0; Most-Recent; Effective; CURRENT

Status: Effective

## 1 Study Objectives and Design

## 1.1 Study Objectives

#### **PRIMARY OBJECTIVE**

The primary objective is to assess initial safety and performance of the soft contact lens when worn in an extended wear modality (ie, up to 6 nights/7 days of continuous wear) as compared to the Biofinity soft contact lens.

#### 1.2 Study Description

Key components of the study are summarized in Table 1-1.

| Table 1 | <b>Study Description Summary</b> |
|---------|----------------------------------|
|---------|----------------------------------|

| Study Design | Prospective, randomized, controlled, double-masked, |
|---|---|
| | contralateral |
| Study Population | Volunteer subjects aged 18 or over who are adapted soft contact |
| | lens wearers, excluding Biofinity habitual wearers, have at least |
| | 3 months of soft contact lens wearing experience, and who wear |
| | their habitual lenses at least 5 days per week and in an extended |
| | wear modality a minimum of 1 night per week. Subjects must |
| | require contact lenses in a power range from -1.00 to -6.00 D. |
| | Pregnant and breastfeeding women are excluded from this study. |
| | Target to complete: 30 |
| | Planned to enroll: ~36 |
| Number of Sites | ~3 (US) |
| Test Product | soft contact lenses (LID018869) |
| Control Product | CooperVision® BIOFINITY® (comfilcon A) soft contact lenses |
| | (Biofinity) |
| Ouration of Treatment Up to 6 nights/7 days of continuous wear | |
| Visits | Visit 1, Day 1: Screening/Baseline/Dispense |
| | Visit 2, Day 2: Next Day Follow-up [≤ 4 hours after awakening] |
| | Visit 3, Day 7: Week 1 Follow-up/Exit [7 days (-1 day) of lens |
| | wear (ideally within 4 hours of awakening)] |

Document: TDOC-0057261 Version: 2.0; Most-Recent; Effective; CURRENT

Status: Effective

#### 1.3 Randomization

A member of the Randomization Programming group at Alcon who is not part of the study team will generate the randomized allocation schedule(s) for study lens sequence assignment. Randomization will be implemented in the Electronic Data Capture (EDC)/randomization integration system.

Subjects will be randomized in a 1:1 ratio to receive treatment with one eye and the other lens in the fellow eye, as indicated below:

Sequence 1: (OD)/Biofinity (OS)

Sequence 2: Biofinity (OD)/

#### 1.4 Masking

This is a double-masked study.



## 2 Analysis Sets

### 2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study. For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed, when applicable, from the corresponding lens sequence at the time of clinical assessment.

# 3 Subject Characteristics and Study Conduct Summaries

Demographic information (age, sex, ethnicity, and race) will be tabulated by lens sequence and overall.

The following tables and listings for study conduct summaries will be presented:

Document: TDOC-0057261 Version: 2.0; Most-Recent; Effective; CURRENT

Status: Effective

- Subject Disposition by Lens Sequence
- Analysis Set by Lens
- Subject Accounting by Lens Sequence
- Listing of Lens Sequence Assignment by Investigator
- Listing of Subjects Discontinued from Study
- Listing of Out-of-Window Visits

#### 4 Effectiveness Analysis Strategy

This study defines one primary endpoint \_\_\_\_\_ The Safety Analysis Set will be used for all effectiveness analyses.

Continuous variables will be summarized using the number of observations, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized with counts and percentages from each category.

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out.

#### 4.1 Effectiveness Endpoints

#### **Primary Endpoint**

The primary endpoint is distance visual acuity (VA) with study lenses, collected in Snellen, for each eye. Conversion will be made to the logMAR scale.



Document: TDOC-0057261

Version: 2.0; Most-Recent; Effective; CURRENT

Status: Effective

Effective Date: 21-Jul-2020

### 4.2 Effectiveness Hypotheses

Alcon - Business Use Only Statistical Analysis Plan

#### **Primary Effectiveness**

No inferences are to be made on the primary effectiveness endpoint; therefore, no hypotheses are formulated.



# 4.3 Statistical Methods for Effectiveness Analyses

## 4.3.1 Primary Effectiveness Analyses

Summary statistics will be provided at each visit (Dispense, Next Day Follow-up, Week 1 Follow-up). Descriptive summary statistics will be displayed with counts and percentages on the Snellen categories, and n, mean, standard deviation, median, minimum, and maximum for the converted logMAR values.

Version: 2.0; Most-Recent; Effective; CURRENT Document: TDOC-0057261 Status: Effective

Alcon - Business Use Only Statistical Analysis Plan

Effective Date: 21-Jul-2020

Alcon - Business Use Only Statistical Analysis Plan Effective Date: 21-Jul-2020 Document: TDOC-0057261 Version: 2.0; Most-Recent; Effective; CURRENT Status: Effective

### 5 Safety Analysis Strategy

### 5.1 Safety Endpoints

The safety endpoints are

- Adverse events (AE)
- Biomicroscopy findings
  - o Limbal hyperemia
  - o Bulbar hyperemia
  - Corneal staining
  - Conjunctival staining
  - o Palpebral conjunctival observations
  - Corneal epithelial edema
  - o Corneal stromal edema
  - Corneal vascularization
  - o Conjunctival compression/indention
  - o Chemosis
  - Corneal infiltrates
  - Other findings
- Device deficiencies

## 5.2 Safety Hypotheses

There are no formal safety hypotheses in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of safety endpoints listed in Section 5.1.

Document: TDOC-0057261 Version: 2.0; Most-Recent; Effective; CURRENT

Status: Effective

#### 5.3 Statistical Methods for Safety Analyses

The analysis set for all safety analyses is defined in Section 2.1. Baseline will be defined as the last measurement prior to exposure to study lenses on Visit 1. Safety variables will be summarized descriptively.

#### **5.3.1** Adverse Events

The applicable definition of an AE is in the study protocol. All AEs occurring from when a subject signs informed consent to when a subject exits the study will be accounted for in the reporting.

Analysis and presentation of pre-treatment AEs will be separated from treatment-emergent AEs occurring during the study period. A pre-treatment AE is an event that occurs after signing informed consent but prior to exposure to study lenses. The period for treatment-emergent AE analysis starts from exposure to study lenses until the subject completes or is discontinued from the study. Each AE will be summarized under the exposed lens based upon the event onset date/time.

Descriptive summaries (counts and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities (MedDRA) Preferred Terms (PT). Serious AEs and significant non-serious ocular AEs will be noted. Additionally, relationship to lens will be identified in all AE tables. Unit of presentation for ocular AEs will be eye and nonocular AEs will be subject.

Individual subject listings will be provided for both pre-treatment and treatment-emergent AEs, where any AE leading to study discontinuation will be indicated.

### 5.3.2 Biomicroscopy Findings

Biomicroscopy assessment will be performed at all study visits. The reporting unit for each biomicroscopy finding will be eye.

A summary of grade category counts and percentages will be presented for each parameter at each scheduled visit. Findings collected during unscheduled visits will be presented in a subject listing. Furthermore, a listing of "Other" slit lamp findings will also be provided.

Additionally, for each biomicroscopy parameter, counts and percentages of eyes that experience an increase of  $\geq 2$  grades from baseline (Visit 1) to any subsequent visit will be presented, together with a supportive listing.

Alcon - Business Use Only Statistical Analysis Plan

Version: 2.0; Most-Recent; Effective; CURRENT

Effective Date: 21-Jul-2020

Status: Effective

**Document:** TDOC-0057261

#### 5.3.3 **Device Deficiencies**

A frequency table showing counts for each treatment-emergent Device Deficiency category will be presented. In addition, listings for treatment-emergent and pre-treatment device deficiencies will be provided,



#### 7 **Sample Size and Power Calculations**

Given the early pilot nature of the study, sample size/power calculation is not relevant.

#### 8 References

Not Applicable.

#### 9 **Revision History**

Revision 1

Document: TDOC-0057261 Version: 2.0; Most-Recent; Effective; CURRENT

Status: Effective

This is the first revision (Version 2.0) of the Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 2.0 of the study protocol.



Table Overview of Study Plan .-2

| Procedure / Assessment | Visit 1, Day 1: Screening/ Baseline/ Dispense | Visit 2, Day 2: Next Day Follow-up ≤ 4 hours after awakening | Visit 3, Day 7: Week 1 Follow-up/Exit ^ 7 days (-1 day) of lens wear (Ideally within 4 hours of awakening) | Unscheduled<br>Visit |
|---|---|---|---|---|
| Informed Consent | X | | | |
| Demographics | X | | | |
| Medical History (including pregnancy*) | X | X | X | X |
| Concomitant Medications | X | X | X | X |
| Inclusion/Exclusion | X | | | |
| Habitual lens information* (brand / manufacturer, power, modality/wear success, habitual lens care brand) | X | | | |
| Biomicroscopy (without study lenses) | X | X | X | X |
| Randomize | X | | | |
| IP Dispense | X | | | (X) |
| VA w/ study lenses (OD, OS, Snellen distance) | X | X | X | (X) |

Procedure / Assessment

Device deficiencies

Exit Form

Visit 3, Day 7:

Week 1 Follow-up/Exit ^

7 days (-1 day) of lens wear

(Ideally within 4 hours of

awakening)

 $\mathbf{X}$ 

 $\mathbf{X}$ 

Visit 2, Day 2:

Next Day Follow-up

≤ 4 hours after

awakening

 $\mathbf{X}$ 

(X)

| AEs | X | X | X | X |
|-----|---|---|---|---|

 $\mathbf{X}$ 

(X)

Visit 1, Day 1:

Screening/ Baseline/ Dispense

^ Any subject who exits early from the study (excluding screen failures) must undergo all procedures outlined in Visit 3, as applicable.

Document: TDOC-0057261 Version: 2.0; Most-Recent; Effective; CURRENT

Status: Effective